CLINICAL TRIAL: NCT04443387
Title: Vitamin D Regulates the Expression of Glucocorticoid Receptors in Blood of Severe Asthmatic Patients
Acronym: VitaminD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dubai Health Authority (Other Government)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Bassam Mahboub, Consultant and Head of department (pulmonary unit), Dubai Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MRC-04/2012_06
Record Dates: First submitted 2020-06-12; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: double blinded randomized study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthmatic low vitamin D on treatment (Active Comparator): asthmatic patient low vitamin D level received treatment for Vitamin D 50000IU weekly
  Interventions: Drug: Vitamin D
- Asthmatic low vitamin D on placepo (Placebo Comparator): asthmatic patient low vitamin D level received placepo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D — A double-blinded, randomized, placebo-controlled study of VitD supplementation on 45 asthmatics with VitD deficiency was performed. Moderate to severe asthmatics between 18 and 65 years of age who had clinician-diagnosed asthma with 25-hydroxyvitamin D3 (25 D3) level less than 20ng/mL at the screening visit were recruited at the Rashid Hospital, Dubai, U.A.E., and the Zayed Military Hospital, Abu Dhabi, U.A.E. Subjects were excluded if they had used any previous VitD supplementation, had any other respiratory diseases or co-morbid conditions or were smokers. According to the American Academy of Family Physicians guidelines, participants received 50, 000 IU of VitD orally or placebo weekly over 8 weeks. Subjects were blinded to treatment and allocated to receive a VitD dose or placebo by the randomization schedule.
  Arms: Asthmatic low vitamin D on treatment
Other: Placebo — A double-blinded, randomized, placebo-controlled study of VitD supplementation on 45 asthmatics with VitD deficiency was performed. Moderate to severe asthmatics between 18 and 65 years of age who had clinician-diagnosed asthma with 25-hydroxyvitamin D3 (25 D3) level less than 20ng/mL at the screening visit were recruited at the Rashid Hospital, Dubai, U.A.E., and the Zayed Military Hospital, Abu Dhabi, U.A.E. Subjects were excluded if they had used any previous VitD supplementation, had any other respiratory diseases or co-morbid conditions or were smokers. According to the American Academy of Family Physicians guidelines, participants received 50, 000 IU of VitD orally or placebo weekly over 8 weeks. Subjects were blinded to treatment and allocated to receive a VitD dose or placebo by the randomization schedule.
  Arms: Asthmatic low vitamin D on placepo

SUMMARY:
Vitamin D (VitD) deficiency is a significant public health concern in many areas around the globe which has been associated with many immune-mediated diseases, including asthma. Severe asthma has been linked with a decreased glucocorticoid receptors (GR) ratio (GR-α/ GR-β ratio), indicating steroid hyporesponsiveness. Using combined in silico and in vivo approaches, aimed to explore the immunomodulatory effect of VitD on asthmatic patients diagnosed with hypovitaminosis D.

DETAILED DESCRIPTION:
Vitamin D (VitD) deficiency is a significant public health concern in many areas around the globe which has been associated with many immune-mediated diseases, including asthma. Severe asthma has been linked with a decreased glucocorticoid receptors (GR) ratio (GR-α/ GR-β ratio), indicating steroid hyporesponsiveness. Using combined in silico and in vivo approaches, the investigators aimed to explore the immunomodulatory effect of VitD on asthmatic patients diagnosed with hypovitaminosis D. Methods: In silico tools were used to identify the regulatory effect of VitD supplementation on GR genes. The investigators measured the expression levels of GR-α and the inactive isoform, GR-β, in the blood of adult asthmatics diagnosed with hypovitaminosis D before and after VitD supplementation. Moreover, the blood levels of inflammatory cytokines associated with asthma severity were determined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* age group between 18 and 65 years
* low level of 25-hydroxyvitamin D3 (25 D3) level less than 20ng/mL

Exclusion Criteria:

* smoker patients
* less than 18 years old
* patient on Vitamin D supplementation already

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
The top Vitamin D regulated pathways in response to Steroids by using Comparative Toxicogenomics Database from thousands of experiments. | 8 weeks
  identify VitD targeted enriched pathways, we analyzed Comparative Toxicogenomics .Enriched Ontology Clustering for the identified genes was performed using the Metascape (a web-based tool used for comprehensive gene list annotation and analysis resource)Database from thousands of experiments.
Asthma Severity effects on VDR and steroid receptors genes by inalyzing expression profile of publicly available datasets (GSE69683) which has a large number of participants and detailed clinical information. | 8 weeks
  analyze the expression profile of publicly available datasets (GSE69683) which has a large number of participants and detailed clinical information.
Examine the up-regulation of GR-α receptor by using supplementation of vitamin D on 45 vitamin D deficient asthmatics | 8 weeks
  by doing double-blinded, randomized, placebo-controlled study was performed to test the effect of VitD supplementation on 45 vitamin D deficient asthmatics.Standard statistical t-tests and one-way ANOVA were performed to test for statistical significance between data groups using GraphPad Prism 8 (GraphPad, San Diego, CA, USA). p < 0.05 was considered significant.
Effects of IL-17 and IL-4 cytokines in asthmatic patients while using Vitamin D supplementation by using ELISA assay | 8 weeks
  by doing double-blinded, randomized, placebo-controlled study was performed to test the effect of VitD supplementation on 45 vitamin D deficient asthmatics. Using qRT-PCR expression of the cytokines
Effects of IL-17 and IL-4 cytokines in asthmatic patients while using Vitamin D supplementation by using ELISA assay | 8 weeks
  by doing double-blinded, randomized, placebo-controlled study was performed to test the effect of VitD supplementation on 45 vitamin D deficient asthmatics.using Bioplex multiplex immunoassay (BioRad, CA,USA) was used to assess the protein expression of the cytokines and by measuring fold change.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT04443387/Prot_SAP_000.pdf